CLINICAL TRIAL: NCT04435301
Title: Acoustic-electric Therapy in Patients With Disorders of Consciousness
Brief Title: Oscillatory Acoustic-electric Stimulation in Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Maastricht University (Other); Zhejiang Mingzhou Brain Rehabilitation Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oscillatory stimulation
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2020-06

CONDITIONS: Consciousness Disorder
Keywords: disorders of consciousness; electric stimulation
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamma modulation effect (Experimental): 40Hz current is applied by a battery-driven current stimulator(NeuroConn, Germany). Two pairs of electrodes are attached to the middle and lower part of the face to stimulate the maxillary nerve (V2) and the mandibular nerve (V3), respectively. 40Hz acoustic stimuli and 40Hz electric stimuli are synchronously applied for 40min/day, for a total of 5 days.
  Interventions: Device: DC-Stimulator, NeuroConn, Germany
- Beta modulation effect (Experimental): 28Hz current is applied by a battery-driven current stimulator. Two pairs of electrodes are attached to the middle and lower part of the face to stimulate the maxillary nerve (V2) and the mandibular nerve (V3). 28Hz acoustic stimuli and 28Hz electric stimuli are synchronously applied for 40min/day, for a total of 5 days.
  Interventions: Device: DC-Stimulator, NeuroConn, Germany
- Sham modulation group (Sham Comparator): Sham stimulation was identical to the 40Hz stimulation, except that the acoustic and electric stimulation were ramped down after 0.5 min to remain turned off for the remaining 39.5 min. Sham stimuli are applied for 40min/day, for a total of 5 days.
  Interventions: Device: DC-Stimulator, NeuroConn, Germany

INTERVENTIONS:
Device: DC-Stimulator, NeuroConn, Germany — Neurostimulation device

SUMMARY:
Altered gamma activity has been observed in several neurological and psychiatric disorders, including a reduction in gamma synchronization in patients with disorders of consciousness. Modulation of gamma oscillations with rhythmic stimulation has been used as a possible therapeutic tool. Hence, we try to use acoustic and electric stimulation at gamma frequency to restore brain oscillation and thereby to improve conscious awareness in patients with disorders of consciousness.

DETAILED DESCRIPTION:
We propose a matched-pair parallel study in patients with disorders of consciousness to investigate whether combined acoustic and trigeminal nerve stimulation can modulate brain oscillations, as measured by electroencephalography (EEG), and whether the brain activity changes are coupled with improvements in consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of disorders of consciousness based on CRS-R
* Time post-injury ranging from one to twelve months
* No history of acquired brain injury or psychiatric or neurological diseases

Exclusion Criteria:

* Not medically stable
* Any contraindication to electric stimulation
* Hearing impairment before brain injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised scores | Day 1-5, Day 11-15
  Coma Recovery Scale-Revised(CRS-R) scores are the gold standard for consciousness. CRS-R consists of 23 items, grouped into 6 sub-scales: auditory, visual, motor, oromotor, communication and arousal. The lowest score on each sub-scale represents reflexive activity; the highest represents behaviors mediated by cognitive input. The total score ranges between 0 (worst) and 23 (best).
Neuropsychological assessment | Day 5 and Day 11
  EEG indicators could be used to assess the conscious level, including gamma oscillations and event-related potentials(P300).
Glasgow Outcome Scale-Extended | 1 year after stimulation
  A widely used index for outcomes after brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Study Director — The First Affiliated Hospital, Zhejiang University
Locations (1):
- First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan S, Wu X, Xie M, Li X, Liu C, Su Y, Chen Y, Wu S, Ma C. Trigeminal nerve stimulation successfully awakened an unconscious patient. Brain Stimul. 2019 Mar-Apr;12(2):361-363. doi: 10.1016/j.brs.2018.11.001. Epub 2018 Nov 3. No abstract available. PMID 30448386